CLINICAL TRIAL: NCT06280326
Title: Effect of Different Materials Used in Orogastric Tube Removal on Skin Condition in Premature Babies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal Investigator, PHD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Orogastric Tube Removal
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Skin Conditions
Keywords: neonatal; skin care; sunflower; preterm; slicone based spray
MeSH Terms: conditions — Premature Birth | interventions — Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunflower Oil Group (Experimental): In the experimental group, patch removal will be performed using sunflower oil instead of silicone-based spray remover, which is the routine of the clinic. In children in the experimental group, the patch that has stuck to the baby's skin and needs to be changed is planned to be removed by applying sunflower oil on the patch.
  Interventions: Other: Sunflower oil
- Control group (Active Comparator): In the clinic, the orogastric catheter is fixed above the lip (mustache area) with a hypoallergenic patch. In cases where the oral gastric catheter needs to be replaced or the adhesive patch needs to be renewed, hypoallergenic patches attached to the skin may cause tape abrasions and scratches on the newborn's skin when removed.Silicone-based spray removers are used to avoid causing injuries.
  In the control group in the study, a silicone-based spray remover was used, which is the routine of the clinic, during the removal of hypoallergenic patches attached to the lip (moustache area) to fix the oragastric catheter.
  Interventions: Other: Slicone based spray

INTERVENTIONS:
Other: Sunflower oil — In the experimental group, patch removal will be performed using sunflower oil.
  Arms: Sunflower Oil Group
Other: Slicone based spray — In the control group, clinical routine procedure will be used to remove the patch (silicone based spray.
  Arms: Control group

SUMMARY:
While medical adhesives provide fixation of devices and catheters in neonatal intensive care, problems such as disruption of skin integrity are frequently encountered when removed. The study aims to compare the effectiveness of sunflower oil and silicone-based remover spray used during the removal of medical adhesives used in oragastric catheter fixation in preterm babies in the Neonatal Intensive Care Unit in preventing skin damage.

DETAILED DESCRIPTION:
Use of materials such as an endotracheal tube, orogastric catheter, nasal cannula, and peripheral vein catheter, which are frequently used in neonatal intensive care.

Medical adhesives are needed for fixing. While medical adhesives provide fixation of devices and catheters in neonatal intensive care, problems such as disruption of skin integrity are frequently encountered when removed. Many materials are being tested and developed in clinics to reduce this risk.Skin barrier products minimize trauma in the removal of medical adhesives by creating a protective layer between the epidermis and the adhesive.

Silicone-based spray removers, one of the skin barrier products, are used in the entire patient population, including newborns.Silicone-based spray removers leave residue on the skin as they evaporate easily. doesn't let go. Since it does not contain alcohol, it does not cause pain. Sunflower oil is a traditional method for premature When used in baby massage applied to babies, it increases the weight gain and height growth of babies and reduces the morbidity rate.The study aims to compare the effectiveness of sunflower oil and silicone-based remover spray used during the removal of medical adhesives used in oragastric catheter fixation in preterm babies in the Neonatal Intensive Care Unit in preventing skin damage.

ELIGIBILITY:
Inclusion Criteria:

* Babies born between 32-36 gestational ages
* Babies admitted to Neonatal Intensive Care
* Babies who have not had medical adhesive tape applied to their lips before
* Babies who do not have any skin diseases
* Noninvasive Mechanical Ventilation or Free Ventilation in the Intensive Care Unit
* Babies who need oxygen
* Babies who do not have any obstacle to inserting an oragastric catheter

Exclusion Criteria:

* Babies followed intubated in care
* Babies with any skin disease
* Babies with a disease that is not suitable for oragastric catheter insertion
* Babies for whom medical adhesive should not be applied on the lips

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-06-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Neonatal Skin Condition Score | immediately after removing the patch of the orogastric tube and 1 hours later.
  It is used to evaluate the skin condition of premature, healthy or sick newborns. The scale consists of three parts, each section has an evaluation section. These sections are respectively; dryness, erythema and disruption of skin integrity/peeling. Each section is scored between 1 and 3 on the scale developed as a three-point Likert scale.
  is taking. The lowest score at the end of the scale is 3 and the highest score is 9. The higher the score, the worse the skin condition.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tural Büyük, PhD, Study Chair — Ondokuz Mayıs University
Locations (1):
- Hatice Uzşen, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahin B, Buyuk ET, Uzsen H, Koyun M, Karal FI. Effect of different materials used in the removal of orogastric catheter adhesive on the skin in premature babies in Turkey. J Pediatr Nurs. 2024 Sep-Oct;78:e117-e123. doi: 10.1016/j.pedn.2024.06.026. Epub 2024 Jul 8. PMID 38971633